CLINICAL TRIAL: NCT03496753
Title: Effect of LED Therapy for the Treatment Nipple Fissures: a Randomized Controlled Trial
Brief Title: Effect of LED Therapy for Treatment Nipple Fissure
Acronym: ELTTNF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Lara Jansiski Motta, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LEDNipple01
Record Dates: First submitted 2018-03-28; First posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Nipple Disorder
Keywords: nipple fissure

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: Statistic analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Led Therapy (Experimental): The following will be the phototherapeutic parameters: total spot area: 1.44 cm²; continuous emission mode; output power: 10 mW; infrared wavelength (880 to 904 nm); fluence: 4 J/cm²; and application time: 10 minutes/session. Sessions will be held three times a week on alternating days for six consecutive weeks, totaling 18 sessions.
  Interventions: Device: Led Therapy
- Control (No Intervention): The control group will receive orientation regarding breast care and adequate breastfeeding techniques. The experimental group will receive the same orientation plus phototherapy sessions using a device developed especially for the treatment of nipple trauma. Both groups will be followed up for six consecutive weeks.

INTERVENTIONS:
Device: Led Therapy — The following will be the phototherapeutic parameters: total spot area: 1.44 cm²; continuous emission mode; output power: 10 mW; infrared wavelength (880 to 904 nm); fluence: 4 J/cm²; and application time: 10 minutes/session. Sessions will be held three times a week on alternating days for six consecutive weeks, totaling 18 sessions.
  Arms: Led Therapy

SUMMARY:
Treatment options for nipple fissures include drug therapy with antifungal and antibiotics, topical applications of lanolin, glycerin gel, creams and lotions, the milk itself, hot compresses and silicone nipple shields. Studies involving a light-emitting diode (LED) therapy have demonstrated anti-inflammatory properties, the enhancement of the wound repair process and the control of pain.

DETAILED DESCRIPTION:
Nipple fissures are the second major cause of the discontinuation of breastfeeding, following a sensation of insufficient milk, which leads to bottle feeding. Poor positioning of the child in relation to the breast, an inadequate frequency or duration of breastfeeding and improper suckling are the main causes of nipple fissure. Discontinuing breastfeeding deprives the infant of essential nutrients and also deprives the mother of certain health benefits. Treatment options for nipple fissures include drug therapy with antifungal and antibiotics, topical applications of lanolin, glycerin gel, creams and lotions, the milk itself, hot compresses and silicone nipple shields. Studies involving a light-emitting diode (LED) therapy have demonstrated anti-inflammatory properties, the enhancement of the wound repair process and the control of pain. As it does not cause discomfort, is relatively inexpensive and may impede the discontinuation of breastfeeding, phototherapy could be a viable option for the treatment of nipple fissures.

The aim of this study is to evaluate LED therapy in treatment of nipple fissures

ELIGIBILITY:
Inclusion Criteria:

1. Nursing mothers aged 18 years or older
2. Diagnosis of nipple fissure and nipple pain with a minimum score of 1 on the Store and Champion scales
3. Having given birth to a healthy, full-term child
4. Performing exclusive breastfeeding
5. Newborn with no oral, palatal or maxillofacial abnormalities
6. Newborn weighing between 2500 and 4000 grams

Exclusion Criteria:

1. History of psychological disorder
2. Presence of mastitis
3. Bacterial or fungal infection in breasts
4. Use of breast pump or plastic nipple

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08-20 (Estimated); Primary Completion 2018-09-20 (Estimated); Study Completion 2019-08-20 (Estimated)

PRIMARY OUTCOMES:
Nipple fissure | 1 week
  Nipple fissure will be evaluate with digital calipers - Black Bull Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Mandaqui Hospital, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No